CLINICAL TRIAL: NCT03447769
Title: A Phase III, Multicenter, Randomized, Double Blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Canakinumab Versus Placebo as Adjuvant Therapy in Adult Subjects With Stages AJCC/UICC v. 8 II -IIIA and IIIB (T>5cm N2) Completely Resected (R0) Non-small Cell Lung Cancer (NSCLC)
Brief Title: Brief Title: Study of Efficacy and Safety of Canakinumab as Adjuvant Therapy in Adult Subjects With Stages AJCC/UICC v. 8 II-IIIA and IIIB (T>5cm N2) Completely Resected Non-small Cell Lung Cancer Acronym: CANOPY-A
Acronym: Canopy-A
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Upon review of the primary analysis results, the benefit-risk was assessed by the Steering Committee Members with the decision that the study will be closed. No new safety signals were observed for canakinumab.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885T2301; 2017-004011-39 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; ACZ885; canakinumab; adjuvant; AJCC/UICC v. 8 stages II-IIIA and IIIB (T>5cm N2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- canakinumab (Experimental): Participants received 200mg of canakinumab subcutaneously every 3 weeks for up to 18 cycles (approximately 54 weeks)
  Interventions: Drug: Canakinumab
- Placebo (Placebo Comparator): Participants received canakinumab placebo subcutaneously every 3 weeks for up to 18 cycles (approximately 54 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canakinumab — 200 mg of canakinumab administered subcutaneously on day 1 of every 21-day cycle for 18 cycles. Canakinumab solution for injection was provided by Novartis as ready-to-use pre-filled syringes to be administered by study personnel.
  Other Names: ACZ885
  Arms: canakinumab
Drug: Placebo — Placebo administered subcutaneously on day 1 of every 21-day cycle for 18 cycles. Placebo solution for injection was provided by Novartis as ready-to-use pre-filled syringes to be administered by study personnel.
  Arms: Placebo

SUMMARY:
The primary purpose of the study was to compare the efficacy and safety of canakinumab versus placebo as adjuvant therapy in adult subjects with stages II -IIIA according to the 8th edition of the American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) and the subset of IIIB (T>5cm N2 disease) completely resected (R0) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This was a phase III, multicenter, randomized, double-blind study to evaluate the efficacy and safety of canakinumab as adjuvant therapy in adult patients with stages AJCC/UICC v.8 II-IIIA and IIIB (T>5 cm N2) completely resected (R0) NSCLC.

Approximately 1500 patients were planned to be randomized 1:1 to canakinumab, 200 mg subcutaneously (s.c.) every 3 weeks or matching placebo s.c. every 3 weeks. Patients were planned to continue their assigned treatment until they completed 18 cycles (cycle= 21 days) or experienced any one of the following: non-small cell lung cancer (NSCLC) disease recurrence as determined by Investigator; unacceptable toxicity that precluded further treatment; treatment discontinuation at the discretion of the Investigator or patient; start of a new antineoplastic therapy; death, or loss to follow-up, whichever occurred first. All patients who discontinued from the study treatment were to be followed up every 12 weeks for survival until the final OS analysis or death, loss to follow-up or withdrawal of consent for survival follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Had completely resected (R0) NSCLC AJCC/UICC v. 8 stage IIA-IIIA and IIIB (N2 disease only) OR had NSCLC Stage IIA-IIIA, IIIB (N2 disease only) and were candidates for complete resection surgery.
* Cisplatin-based chemotherapy was mandatory for all subjects (Exception: In subjects with stage IIA disease with no nodal involvement, cisplatin-based chemotherapy could be administered if recommended by the treating physician). When required, a minimum of two cycles of cisplatin-based chemotherapy was mandatory, after which additional therapies could be given based upon local clinical practice and/or guidelines. Typically, chemotherapy was initiated within 60 days of surgery.
* Radiation therapy was allowed if indicated as per local guidelines or practice.
* Had recovered from all toxicities related to prior systemic therapy to grade ≤ 1 (CTCAE v 5.0). Exception to this criterion: subjects with any grade of alopecia and grade 2 or less neuropathy were allowed to enter the study
* Had ECOG performance status (PS) of 0 or 1

Key Exclusion Criteria:

* Had unresectable or metastatic disease, positive microscopic margins on the pathology report, and/or gross disease remaining at the time of surgery
* Had received any neoadjuvant therapy
* Had presence or history of a malignant disease, other than the resected NSCLC, that had been diagnosed and/or required therapy within the past 3 years Exceptions to this exclusion included the following: completely resected basal cell and squamous cell skin cancers, completely resected carcinoma in situ of any type and hormonal maintenance for breast and prostate cancer > 3 years.
* Had a history of current diagnosis of cardiac disease
* Had uncontrolled diabetes
* Had known active or recurrent hepatic disorder including cirrhosis, hepatitis B and C (positive or indeterminate central laboratory results)
* Subjects had to be evaluated for tuberculosis as per local treatment guidelines or clinical practice. Subjects with active tuberculosis were not eligible.
* Had suspected or proven immunocompromised state as described in the protocol
* Had live and attenuated vaccination within 3 months prior to first dose of study drug (e.g. MMR, Yellow Fever, Rotavirus, Smallpox, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1382 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (251):
- United States (21):
  - Highlands Oncology Group ., Fayetteville, Arkansas
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - University of California at Los Angeles, Los Angeles, California
  - VA Palo Alto Health Care System CRLX030A2301, Palo Alto, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers Denver-Mdtn(Bone&MarrowTransp), Longmont, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Advanced Medical Specialties Drug Ship - 2, Miami, Florida
  - Florida Cancer Affiliates of Ocala, Ocala, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Rush University Medical Center Regulatory, Chicago, Illinois
  - Cancer Center of Kansas Dept.ofCancerCtr.ofKansas, Wichita, Kansas
  - VA Nebraska-W IA Health Care System ., Omaha, Nebraska
  - Louis Stokes Cleveland Department of Veterans Affairs MC ., Cleveland, Ohio
  - Oncology Associates of Oregon, PC, Eugene, Oregon
  - Chattanooga Oncology and Hematology Associates PC Chattanooga Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology MamieMcFaddenWardCtr, Dallas, Texas
  - Virginia Cancer Specialists Fairfax Northern Virginia, Fairfax, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc ., Salem, Virginia
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, Córdoba
- Austria (4):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Klagenfurt
  - Novartis Investigative Site, Krems
  - Novartis Investigative Site, Vienna
- Brazil (4):
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Teresina, Piauí
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Novartis Investigative Site, Santiago, Chile
- China (23):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Zhanjing, Guangong
  - Novartis Investigative Site, Zunyi, Guizhou
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Jinan, Shandong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Shenyang, Shengyang
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Changsha
  - Novartis Investigative Site, Chengdu
  - Novartis Investigative Site, Fujian
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Bogotá, Colombia
- Czechia (2):
  - Novartis Investigative Site, Ostrava Vitkovice
  - Novartis Investigative Site, Prague
- France (21):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Le Mans, Cedex 09
  - Novartis Investigative Site, Montpellier, Herault
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, La Rochelle
  - Novartis Investigative Site, La Seyne-sur-Mer
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Suresnes
  - Novartis Investigative Site, Toulouse
- Georgia (2):
  - Novartis Investigative Site, Batumi
  - Novartis Investigative Site, Tbilisi
- Germany (23):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Gauting, Bavaria
  - Novartis Investigative Site, Bochum, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Solingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Athens, Attica
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
  - Novartis Investigative Site, Tuenmen
- Hungary (2):
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Reykjavik, Iceland
- India (4):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Delhi
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Holon
- Italy (11):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
- Japan (23):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Hirosaki, Aomori
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Iizuka, Fukuoka
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Shiwa-gun, Iwate
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Natori-shi, Miyagi
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Sunto Gun, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Ube, Yamaguchi
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Wakayama
- Novartis Investigative Site, Amman, Jordan
- Lebanon (4):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
  - Novartis Investigative Site, Tripoli
- Malaysia (3):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Pulau Pinang
- Norway (4):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Drammen
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Tromsø
- Novartis Investigative Site, Panama City, Panama
- Peru (2):
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
- Novartis Investigative Site, Makati City, Philippines
- Poland (6):
  - Novartis Investigative Site, Krakow, Ma3opolska
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Olsztyn
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Porto
- Romania (4):
  - Novartis Investigative Site, Floreşti, Cluj
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Iași
- Russia (9):
  - Novartis Investigative Site, Arkhangelsk
  - Novartis Investigative Site, Kaliningrad
  - Novartis Investigative Site, Moscow Region Istra Village
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Pushkin Saint Petersburg
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- Novartis Investigative Site, Ljubljana, Slovenia
- South Korea (5):
  - Novartis Investigative Site, Jeollanam-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Geneva
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Hualien City
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (4):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chaingmai
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Pendik Istanbul, Turkey
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (14):
  - Novartis Investigative Site, Cambridge, Cambrigdeshire
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Cheltenham, Gloucestershire
  - Novartis Investigative Site, Metropolitan Borough of Wirral, Merseyside
  - Novartis Investigative Site, Ipswich, Suffolk
  - Novartis Investigative Site, Guildford, Surrey
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Stoke-on-Trent
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data will be available according to the process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Garon EB, Lu S, Goto Y, De Marchi P, Paz-Ares L, Spigel DR, Thomas M, Yang JC, Ardizzoni A, Barlesi F, Orlov S, Yoshioka H, Mountzios G, Khanna S, Bossen C, Carbini M, Turri S, Myers A, Cho BC. Canakinumab as Adjuvant Therapy in Patients With Completely Resected Non-Small-Cell Lung Cancer: Results From the CANOPY-A Double-Blind, Randomized Clinical Trial. J Clin Oncol. 2024 Jan 10;42(2):180-191. doi: 10.1200/JCO.23.00910. Epub 2023 Oct 3. PMID 37788412
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1875

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 290 centers in 41 countries. A total of 1830 subjects were screened of which 1382 participants were randomized to treatment on a 1:1 basis.
Pre-assignment Details: 1 participant randomized in the canakinumab arm was never treated due to subject decision.
  The numbers in the patient disposition table correspond to the treatment period.
Groups:
- Canakinumab: Participants receive 200mg of canakinumab subcutaneously every 3 weeks for up to 18 cycles (approximately 54 weeks)
- Placebo: Participants receive canakinumab placebo subcutaneously every 3 weeks for up to 18 cycles (approximately 54 weeks)
Period: Overall Study
Arm/Group | Canakinumab | Placebo
Started | 693 | 689
Treated | 692 | 689
Completed (Participants who completed treatment) | 414 | 420
Not Completed | 279 | 269
Not completed — Progressive disease | 138 | 148
Not completed — Study terminated by Sponsor | 60 | 44
Not completed — Adverse Event | 34 | 31
Not completed — Patient decision | 27 | 27
Not completed — Protocol deviation | 4 | 6
Not completed — Death | 2 | 7
Not completed — Technical problems | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canakinumab | Placebo | Total
Number analyzed (Participants) | 693 | 689 | 1382
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (8.90) | 61.6 (9.00) | 61.6 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 257 | 520
  Male | 430 | 432 | 862
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 393 | 391 | 784
  Asian | 248 | 236 | 484
  Black or African American | 3 | 4 | 7
  American Indian or Alaska Native | 0 | 5 | 5
  Multiple | 0 | 1 | 1
  Missing | 49 | 52 | 101

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS) by Local Investigator
Description: DFS is the time from the date of randomization to the date of the first documented NSCLC disease recurrence as assessed by local investigator radiologically or death due to any cause. Disease recurrence included diagnoses of new primary lung malignancies. Clinical deterioration was not considered as a recurrence of disease. In case of non-conclusive radiological evidence, a biopsy assessment was performed to confirm NSCLC recurrence.
  The median DFS was estimated using the Kaplan-Meier method. DFS was censored if no DFS event was observed prior to the analysis cut-off date or subjects who received any subsequent anti-neoplastic therapy for NSCLC. The censoring date was the date of last assessment before the cut-off date or NSCLC related anti-neoplastic therapy date.
Time Frame: Up to approximately 4 years
Population: Full Analysis Set (FAS) including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months | 35.02 [28.55 to NA] — NA: Not estimable due to the insufficient number of participants with events | 29.73 [23.72 to NA] — NA: Not estimable due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; Test type: Superiority; p = 0.258, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.14] — The HR for DFS was calculated, along with its 95% confidence interval, from a stratified Cox model using the same stratification factors as those for the log-rank test

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is the time from the date of randomization to the date of death due to any cause. The OS was censored at the latest date the subject was known to be alive. The OS distribution was estimated using the Kaplan-Meier method, and Kaplan-Meier medians and 95% confidence intervals of the medians were presented for each treatment group.
Time Frame: Up to approximately 4.3 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months | 51.12 [46.95 to NA] — NA = Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA = Not estimable due to the insufficient number of participants with events

3. Secondary Outcome: Overall Survival (OS) in PD-L1 Subgroups
Description: Overall Survival (OS) is the time from the date of randomization to the date of death due to any cause. The OS was censored at the latest date the subject was known to be alive. The OS distribution was estimated using the Kaplan-Meier method, and Kaplan-Meier curves, medians and 95% confidence intervals of the medians were presented for each treatment group. OS analysis was performed by programmed cell death-ligand 1 (PD-L1) expression status: PD-L1 <1%, PD-L1 ≥1% and <49%, and PD-L1 ≥50%.
Time Frame: Up to approximately 4.3 years
Population: Participants to whom study treatment was assigned by randomization with a valid baseline measurement of PD-L1 expression.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 396 | 418
Months
  PD-L1 <1%: number analyzed (Participants) | 211 | 203
  PD-L1 <1% | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events
  PD-L1 ≥1% and <49%: number analyzed (Participants) | 99 | 119
  PD-L1 ≥1% and <49% | 46.95 [22.11 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events
  PD-L1 ≥50%: number analyzed (Participants) | 86 | 96
  PD-L1 ≥50% | 51.12 [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events

4. Secondary Outcome: Overall Survival (OS) in CD8 Subgroups
Description: Overall Survival (OS) is the time from the date of randomization to the date of death due to any cause. The OS was censored at the latest date the subject was known to be alive. The OS distribution was estimated using the Kaplan-Meier method, and Kaplan-Meier medians and 95% confidence intervals of the medians were presented for each treatment group. OS analysis was performed by CD8 subgroups with the median of baseline CD8 expression as cut-off.
Time Frame: up to approximately 4.3 years
Population: Participants to whom study treatment was assigned by randomization with a valid baseline measurement of CD8 expression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 429 | 449
Months
  CD8 < median: number analyzed (Participants) | 213 | 225
  CD8 < median | 46.95 [32.23 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events
  CD8 ≥ median: number analyzed (Participants) | 216 | 224
  CD8 ≥ median | 51.12 [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events

5. Secondary Outcome: Lung Cancer Specific Survival (LCSS)
Description: LCSS is defined as the time from date of randomization to the date of death due to lung cancer. The LCSS distribution was estimated using the Kaplan-Meier method, and Kaplan-Meier medians and 95% confidence intervals of the medians were presented for each treatment group.
Time Frame: Up to approximately 4.3 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months | 51.12 [44.71 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events

6. Secondary Outcome: Disease Free Survival (DFS) by Local Investigator in PD-L1 Subgroups
Description: DFS is the time from the date of randomization to the date of the first documented NSCLC disease recurrence as assessed by local investigator radiologically or death due to any cause. Disease recurrence included diagnoses of new primary lung malignancies. Clinical deterioration was not considered as a recurrence of disease. In case of non-conclusive radiological evidence, a biopsy assessment was performed to confirm NSCLC recurrence.
  The median DFS was estimated using the Kaplan-Meier method. DFS was censored if no DFS event was observed prior to the analysis cut-off date or subjects who received any subsequent anti-neoplastic therapy for NSCLC. The censoring date was the date of last assessment before the cut-off date or NSCLC related anti-neoplastic therapy date.
  DFS analysis was performed by baseline programmed cell death-ligand 1 (PD-L1) expression status: PD-L1 <1%, PD-L1 ≥1% and <49%, and PD-L1 ≥50%.
Time Frame: Up to approximately 4 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 396 | 418
Months
  PD-L1 <1%: number analyzed (Participants) | 211 | 203
  PD-L1 <1% | 30.72 [23.52 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [23.03 to NA] — NA: Not estimable due to the insufficient number of participants with events
  PD-L1 ≥1% and <49%: number analyzed (Participants) | 99 | 119
  PD-L1 ≥1% and <49% | 30.42 [21.42 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [17.05 to NA] — NA: Not estimable due to the insufficient number of participants with events
  PD-L1 ≥50%: number analyzed (Participants) | 86 | 96
  PD-L1 ≥50% | 46.95 [19.45 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [22.31 to NA] — NA: Not estimable due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; PD-L1 <1%; Test type: Superiority; p = 0.676, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.76 to 1.58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Canakinumab vs Placebo; PD-L1 ≥1% and <49%; Test type: Superiority; p = 0.036, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.34 to 1.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Canakinumab vs Placebo; PD-L1 ≥50%; Test type: Superiority; p = 0.823, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.73 to 2.43] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Disease Free Survival (DFS) by Local Investigator in CD8 Subgroups
Description: DFS is the time from the date of randomization to the date of the first documented NSCLC disease recurrence as assessed by local investigator radiologically or death due to any cause. Disease recurrence included diagnoses of new primary lung malignancies. Clinical deterioration was not considered as a recurrence of disease. In case of non-conclusive radiological evidence, a biopsy assessment was performed to confirm NSCLC recurrence.
  The median DFS was estimated using the Kaplan-Meier method. DFS was censored if no DFS event was observed prior to the analysis cut-off date or subjects who received any subsequent anti-neoplastic therapy for NSCLC. The censoring date was the date of last assessment before the cut-off date or NSCLC related anti-neoplastic therapy date.
  DFS analysis was performed by CD8 subgroups with the median of baseline CD8 expression as cut-off.
Time Frame: Up to approximately 4 years
Population: Participants to whom study treatment was assigned by randomization with a valid baseline measurement of CD8 expression
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 429 | 449
Months
  CD8 < median: number analyzed (Participants) | 213 | 225
  CD8 < median | 26.58 [20.67 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [25.03 to NA] — NA: Not estimable due to the insufficient number of participants with events
  CD8 ≥ median: number analyzed (Participants) | 216 | 224
  CD8 ≥ median | 46.95 [28.81 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [23.89 to NA] — NA: Not estimable due to the insufficient number of participants with events
Statistical Analysis 1: Comparison: Canakinumab vs Placebo; CD8 < median; Test type: Superiority; p = 0.872, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.87 to 1.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Canakinumab vs Placebo; CD8 ≥ median; Test type: Superiority; p = 0.303, Stratified log-rank test — 1-sided p-value; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.62 to 1.33] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Canakinumab Serum Concentrations
Description: Serum concentrations of canakinumab were determinded using an ELISA method.
Time Frame: Cycle 1 on day 1 (pre-dose), day 8 and 15; Cycle 2, 4, 6, 9 and 12 on day 1 (pre-dose). Cycle=21 days
Population: The Pharmacokinetic analysis set (PAS) including all subjects who received at least one dose of canakinumab and provided at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Canakinumab
Number analyzed (Participants) | 664
ug/ml
  Cycle 1 Day 1 | 0 (0)
  Cycle 1 Day 8: number analyzed (Participants) | 569
  Cycle 1 Day 8 | 18.1 (6.53)
  Cycle 1 Day 15: number analyzed (Participants) | 611
  Cycle 1 Day 15 | 16.9 (5.43)
  Cycle 2 Day 1: number analyzed (Participants) | 636
  Cycle 2 Day 1 | 15.0 (4.91)
  Cycle 4 Day 1: number analyzed (Participants) | 611
  Cycle 4 Day 1 | 29.7 (10.3)
  Cycle 6 Day 1: number analyzed (Participants) | 559
  Cycle 6 Day 1 | 34.7 (13.0)
  Cycle 9 Day 1: number analyzed (Participants) | 530
  Cycle 9 Day 1 | 37.1 (14.5)
  Cycle 12 Day 1: number analyzed (Participants) | 502
  Cycle 12 Day 1 | 38.6 (15.5)

9. Secondary Outcome: Canakinumab Anti-drug Antibody (ADA) Prevalence at Baseline
Description: Canakinumab ADA prevalence at baseline was calculated as the percentage of participants who had an ADA positive result at baseline
Time Frame: Baseline
Population: All subjects who received at least one dose of canakinumab
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 692
Participants | 8

10. Secondary Outcome: Canakinumab ADA Incidence
Description: Canakinumab ADA incidence on-treatment was calculated as the percentage of participants who were treatment-induced ADA positive (post-baseline ADA positive with ADA-negative sample at baseline) and treatment-boosted ADA positive (post-baseline ADA positive with titer that was at least the fold titer change greater than the ADA-positive baseline titer)
Time Frame: From baseline up to 130 days after end of treatment, assessed up to approx. 1.5 years
Population: All subjects who received at least one dose of canakinumab
Measure: Count of Participants; unit: Participants
Arm/Group | Canakinumab
Number analyzed (Participants) | 692
Participants | 7

11. Secondary Outcome: Time to Definitive 10 Point Deterioration Symptom Scores of Pain,Cough and Dyspnea Per European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ)- Lung Cancer (LC) 13 Questionnaire
Description: The Lung Cancer module of the EORTC's quality of life questionnaire (EORTC QLQ-LC13) was used in conjunction with the EORTC QLQ-C30 and provided information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporated one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores ranged from 0 to 100. A high score indicated a high level of symptoms.
  The time to definitive 10 point deterioration symptom scores of pain, cough and dyspnea was defined as the time from the date of randomization to the date of event, which was defined as at least 10 points relative to baseline worsening of the EORTC QLQ-LC13 symptom score with no later change below this threshold or death due to any cause, whichever occurred earlier.
Time Frame: From baseline up to approximately 4 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months
  Pain | NA [35.45 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events
  Cough | NA [35.06 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [34.99 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Dyspnea | 28.88 [23.10 to 34.96] | 34.99 [23.13 to NA] — NA: Not estimable due to the insufficient number of participants with events

12. Secondary Outcome: Time to Definitive 10 Point Deterioration of Global Health Status/Quality of Life (QoL), Shortness of Breath and Pain Per EORTC QLQ-C30 Questionnaire
Description: The EORTC QLQ-C30 was a questionnaire developed to assess the health-related quality of life of cancer participants. It assessed 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/QoL scale. All domain scores ranged from 0 to 100. A high score for the functional or global health status scales indicated a high level of functioning or QoL; a high score for a symptom scale indicated a high level of symptoms.
  The time to definitive 10 point deterioration of global health status/QoL, shortness of breath and pain was defined as the time from the date of randomization to the date of event, which was defined as at least 10 points relative to baseline worsening of the EORTC QLQ-C30 score with no later change below this threshold or death due to any cause, whichever occured earlier.
Time Frame: From baseline up to approximately 4 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months
  Global health status/QoL | 34.99 [29.93 to NA] — NA: Not estimable due to the insufficient number of participants with events | 35.15 [35.15 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Shortness of breath | NA [NA to NA] — NA: Not estimable due to the insufficient number of participants with events | 35.15 [34.99 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Pain | 29.93 [28.29 to 35.22] | 36.44 [34.99 to NA] — NA: Not estimable due to the insufficient number of participants with events

13. Secondary Outcome: Time to First 10 Point Deterioration for Symptom Scores of Pain, Cough and Dyspnea Per EORTC QLQ-LC13 Questionnaire
Description: The Lung Cancer module of the EORTC's quality of life questionnaire (EORTC QLQ-LC13) was used in conjunction with the EORTC QLQ-C30 and provided information on an additional 13 items specifically related to lung cancer. The lung cancer module incorporated one multi-item scale to assess dyspnea, and 9 single items assessing pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All of the domain scores ranged from 0 to 100. A high score indicated a high level of symptoms.
  The time to first 10 point deterioration symptom scores of pain, cough and dyspnea was defined as the time from the date of randomization to the first onset of at least 10 points absolute increase from baseline (worsening) in symptoms scores or death due to any cause, whichever occurred earlier.
Time Frame: From baseline up to approximately 4 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months
  Pain | 35.15 [26.58 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [23.06 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Cough | 15.44 [10.38 to 23.06] | 15.01 [9.69 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Dyspnea | 4.17 [3.42 to 5.55] | 4.86 [3.48 to 6.97]

14. Secondary Outcome: Time to First 10 Point Deterioration of Global Health Status/QoL, Shortness of Breath and Pain Per EORTC QLQ-C30 Questionnaire
Description: The EORTC QLQ-C30 was a questionnaire developed to assess the health-related quality of life of cancer participants. It assessed 15 domains consisting of 5 functional domains (physical, role, emotional, cognitive, social) and 9 symptom domains (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties) and a global health status/QoL scale. All domain scores ranged from 0 to 100. A high score for the functional or global health status scales indicated a high level of functioning or QoL; a high score for a symptom scale indicated a high level of symptoms.
  The time to first 10 point deterioration of global health status/QoL, shortness of breath and pain scores was defined as the time from the date of randomization to the first onset of at least 10 points absolute increase from baseline (worsening) in symptoms scores or death due to any cause, whichever occurred earlier.
Time Frame: From baseline up to approximately 4 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Months
  Global health status/QoL | 9.23 [7.10 to 11.76] | 9.07 [7.62 to 11.76]
  Shortness of breath | 29.14 [23.03 to NA] — NA: Not estimable due to the insufficient number of participants with events | NA [23.13 to NA] — NA: Not estimable due to the insufficient number of participants with events
  Pain | 5.49 [4.21 to 6.90] | 5.62 [4.17 to 7.62]

15. Secondary Outcome: Change From Baseline in the Utility Score of the EuroQoL- 5 Dimension- 5 Level (EQ-5D-5L)
Description: EQ-5D-5L was a standardized questionnaire that measured health-related QoL. EQ-5D-5L consisted of 2 components: a health state profile and a visual analogue scale. The health state profile included five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels ranging from 1 (no problems) to 5 (extreme problems).
  The EQ-5D-5L health state profile responses were converted into single index utility score, ranging from -1 to 1, where lower scores representing a higher level of dysfunction. Published weights are available enabling the calculation of the utility score. A positive change from baseline indicated improvement. This endpoint was assessed throughout the study, including safety and efficacy follow-up (FU) visits. Safety FU visits: every 4 weeks after end of treatment up to 130 days post-last dose. Efficacy FU visits: at 18, 24, 30, 36 and 48 months post-randomization (if no recurrence observed during treatment or safety FU)
Time Frame: Baseline, every 3 weeks for 14 months; end of treatment; every 4 weeks up to 130 days post-treatment; at 18,24,30,36 and 48 months post-randomization (if no recurrence); 7 and 28 days post-disease progression, up to approx. 4 years.
Population: All participants to whom study treatment was assigned by randomization with data available at the specified time points. Number analyzed refers to the number of participants with an evaluable value at the specified time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 643 | 629
Score on a scale
  Week 3 | 0.0 (0.11) | 0.0 (0.12)
  Week 6: number analyzed (Participants) | 626 | 614
  Week 6 | 0.0 (0.13) | 0.0 (0.12)
  Week 9: number analyzed (Participants) | 619 | 603
  Week 9 | 0.0 (0.13) | 0.0 (0.13)
  Week 12: number analyzed (Participants) | 619 | 604
  Week 12 | 0.0 (0.12) | 0.0 (0.12)
  Week 15: number analyzed (Participants) | 581 | 572
  Week 15 | 0.0 (0.13) | 0.0 (0.12)
  Week 18: number analyzed (Participants) | 564 | 558
  Week 18 | 0.0 (0.13) | 0.0 (0.13)
  Week 21: number analyzed (Participants) | 555 | 556
  Week 21 | 0.0 (0.13) | 0.0 (0.15)
  Week 24: number analyzed (Participants) | 551 | 550
  Week 24 | 0.0 (0.14) | 0.0 (0.14)
  Week 27: number analyzed (Participants) | 528 | 532
  Week 27 | 0.0 (0.13) | 0.0 (0.14)
  Week 30: number analyzed (Participants) | 523 | 504
  Week 30 | 0.0 (0.13) | 0.0 (0.14)
  Week 33: number analyzed (Participants) | 509 | 506
  Week 33 | 0.0 (0.13) | 0.0 (0.14)
  Week 36: number analyzed (Participants) | 502 | 502
  Week 36 | 0.0 (0.14) | 0.0 (0.15)
  Week 39: number analyzed (Participants) | 461 | 471
  Week 39 | 0.0 (0.15) | 0.0 (0.13)
  Week 42: number analyzed (Participants) | 451 | 452
  Week 42 | 0.0 (0.15) | 0.0 (0.14)
  Week 45: number analyzed (Participants) | 440 | 428
  Week 45 | 0.0 (0.14) | 0.0 (0.14)
  Week 48: number analyzed (Participants) | 423 | 422
  Week 48 | 0.0 (0.14) | 0.0 (0.15)
  Week 51: number analyzed (Participants) | 385 | 406
  Week 51 | 0.0 (0.13) | 0.0 (0.14)
  Week 54: number analyzed (Participants) | 17 | 11
  Week 54 | 0.0 (0.18) | 0.1 (0.12)
  Week 57: number analyzed (Participants) | 1 | 1
  Week 57 | 0.0 | -0.1
  Week 60: number analyzed (Participants) | 1 | 1
  Week 60 | -0.2 | -0.1
  Week 63: number analyzed (Participants) | 1 | 0
  Week 63 | 0.0 |
  Week 69: number analyzed (Participants) | 1 | 0
  Week 69 | 0.0 |
  Safety FU 1: number analyzed (Participants) | 431 | 443
  Safety FU 1 | 0.0 (0.15) | 0.0 (0.14)
  Safety FU 2: number analyzed (Participants) | 421 | 432
  Safety FU 2 | 0.0 (0.14) | 0.0 (0.14)
  Safety FU 3: number analyzed (Participants) | 420 | 418
  Safety FU 3 | 0.0 (0.14) | 0.0 (0.15)
  Safety FU 4: number analyzed (Participants) | 392 | 406
  Safety FU 4 | 0.0 (0.15) | 0.0 (0.16)
  Safety FU 5: number analyzed (Participants) | 392 | 397
  Safety FU 5 | 0.0 (0.15) | 0.0 (0.14)
  Efficacy FU 1: number analyzed (Participants) | 237 | 254
  Efficacy FU 1 | 0.0 (0.16) | 0.0 (0.14)
  Efficacy FU 2: number analyzed (Participants) | 179 | 178
  Efficacy FU 2 | 0.0 (0.15) | 0.0 (0.16)
  Efficacy FU 3: number analyzed (Participants) | 124 | 116
  Efficacy FU 3 | 0.0 (0.14) | 0.0 (0.15)
  Efficacy FU 4: number analyzed (Participants) | 67 | 72
  Efficacy FU 4 | 0.0 (0.13) | 0.0 (0.15)
  Efficacy FU 5: number analyzed (Participants) | 15 | 7
  Efficacy FU 5 | 0.0 (0.10) | -0.1 (0.17)
  7 days post disease progression: number analyzed (Participants) | 29 | 22
  7 days post disease progression | -0.1 (0.16) | -0.1 (0.22)
  28 days post disease progression: number analyzed (Participants) | 86 | 79
  28 days post disease progression | -0.1 (0.18) | -0.1 (0.18)

16. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from day of participant's informed consent to the day before first dose of study medication.
  On-treatment deaths were collected from start of treatment to 130 days after last dose.
  Post-treatment follow-up deaths were collected from day 131 after last dose of study treatment to end of study.
Time Frame: Pre-treatment: Up to 28 days prior to treatment. On-treatment: Up to approx. 1.5 years. Post-treatment follow-up: Up to approx. 4.3 years
Population: FAS including all participants to whom study treatment was assigned by randomization
Measure: Number; unit: Participants
Arm/Group | Canakinumab | Placebo
Number analyzed (Participants) | 693 | 689
Participants
  Pre-treatment deaths | 0 | 0
  On-treatment deaths: number analyzed (Participants) | 692 | 689
  On-treatment deaths | 9 | 17
  Post-treatment follow-up deaths: number analyzed (Participants) | 671 | 662
  Post-treatment follow-up deaths | 53 | 51
  All deaths | 62 | 68

ADVERSE EVENTS:
Time Frame: Pre-treatment: from study consent to the day before first dose, up to 28 days. On-treatment: from first dose of study treatment to 130 days after last dose of study medication, up to approx. 1.5 years. Post-treatment follow-up: from 131 days after last dose of study medication until the end of the study, up to approx. 4.3 years.
Description: Treatment-emergent AEs refer to any signs or symptoms observed during the study treatment and up to 130 days after treatment, considering the Safety Set (including participants who received at least one dose of study treatment). All-Cause Mortality analysis encompasses the Full Analysis Set, including all participants to whom study treatment was assigned by randomization
Groups:
- All Participants - Pre-treatment: Deaths collected in the pre-treatment period (from day of patient's informed consent to the day before first administration of study treatment)
- Canakinumab - On-treatment; Placebo - On-treatment: AEs collected during on-treatment period (up to 130 days post-treatment)
- Canakinumab - Post-treatment Follow-up: Deaths collected in the post-treatment follow-up period (starting from day 131 post- treatment). No AEs were collected during this period
- Placebo - Post-treatment Follow-up: Deaths collected in the post-treatment follow-up period (starting from day 131 post-treatment). No AEs were collected during this period
Arm/Group | All Participants - Pre-treatment | Canakinumab - On-treatment | Canakinumab - Post-treatment Follow-up | Placebo - On-treatment | Placebo - Post-treatment Follow-up
All-Cause Mortality (participants affected / at risk) | 0/1382 | 9/692 | 53/671 | 17/689 | 51/662
Serious Adverse Events (participants affected / at risk) | 0/0 | 141/692 | 0/0 | 146/689 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 465/692 | 0/0 | 455/689 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants - Pre-treatment (N=0) | Canakinumab - On-treatment (N=692) | Canakinumab - Post-treatment Follow-up (N=0) | Placebo - On-treatment (N=689) | Placebo - Post-treatment Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | 0 | NA | 1 | NA
Thrombocytosis (Blood and lymphatic system disorders) | NA | 0 | NA | 1 | NA
Acute coronary syndrome (Cardiac disorders) | NA | 0 | NA | 1 | NA
Acute myocardial infarction (Cardiac disorders) | NA | 0 | NA | 1 | NA
Angina pectoris (Cardiac disorders) | NA | 3 | NA | 2 | NA
Atrial fibrillation (Cardiac disorders) | NA | 2 | NA | 0 | NA
Atrial flutter (Cardiac disorders) | NA | 0 | NA | 1 | NA
Cardiac arrest (Cardiac disorders) | NA | 1 | NA | 0 | NA
Cardiac failure (Cardiac disorders) | NA | 0 | NA | 1 | NA
Cardiac failure congestive (Cardiac disorders) | NA | 1 | NA | 0 | NA
Cardiac ventricular thrombosis (Cardiac disorders) | NA | 0 | NA | 1 | NA
Cardiovascular insufficiency (Cardiac disorders) | NA | 0 | NA | 1 | NA
Coronary artery disease (Cardiac disorders) | NA | 1 | NA | 1 | NA
Myocardial infarction (Cardiac disorders) | NA | 1 | NA | 4 | NA
Myocardial ischaemia (Cardiac disorders) | NA | 0 | NA | 2 | NA
Pericarditis constrictive (Cardiac disorders) | NA | 0 | NA | 1 | NA
Supraventricular tachycardia (Cardiac disorders) | NA | 1 | NA | 0 | NA
Vertigo (Ear and labyrinth disorders) | NA | 0 | NA | 1 | NA
Retinal detachment (Eye disorders) | NA | 0 | NA | 1 | NA
Retinal tear (Eye disorders) | NA | 0 | NA | 1 | NA
Rhegmatogenous retinal detachment (Eye disorders) | NA | 1 | NA | 0 | NA
Abdominal hernia (Gastrointestinal disorders) | NA | 1 | NA | 0 | NA
Abdominal pain (Gastrointestinal disorders) | NA | 3 | NA | 2 | NA
Colitis (Gastrointestinal disorders) | NA | 1 | NA | 0 | NA
Constipation (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA
Diarrhoea (Gastrointestinal disorders) | NA | 1 | NA | 1 | NA
Enterocolitis (Gastrointestinal disorders) | NA | 1 | NA | 0 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | NA | 1 | NA | 2 | NA
Gastrointestinal pain (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA
Haemorrhoids (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA
Large intestine polyp (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA
Lumbar hernia (Gastrointestinal disorders) | NA | 1 | NA | 0 | NA
Pancreatic cyst (Gastrointestinal disorders) | NA | 1 | NA | 0 | NA
Pancreatitis acute (Gastrointestinal disorders) | NA | 1 | NA | 1 | NA
Rectal haemorrhage (Gastrointestinal disorders) | NA | 0 | NA | 1 | NA
Vomiting (Gastrointestinal disorders) | NA | 1 | NA | 1 | NA
Asthenia (General disorders) | NA | 1 | NA | 1 | NA
Chest pain (General disorders) | NA | 0 | NA | 2 | NA
Fatigue (General disorders) | NA | 0 | NA | 1 | NA
Non-cardiac chest pain (General disorders) | NA | 2 | NA | 2 | NA
Pain (General disorders) | NA | 0 | NA | 1 | NA
Pyrexia (General disorders) | NA | 2 | NA | 1 | NA
Biliary colic (Hepatobiliary disorders) | NA | 0 | NA | 1 | NA
Cholecystitis (Hepatobiliary disorders) | NA | 1 | NA | 3 | NA
Cholelithiasis (Hepatobiliary disorders) | NA | 0 | NA | 1 | NA
Gallbladder obstruction (Hepatobiliary disorders) | NA | 1 | NA | 0 | NA
Hepatitis acute (Hepatobiliary disorders) | NA | 1 | NA | 0 | NA
Appendicitis (Infections and infestations) | NA | 0 | NA | 1 | NA
Asymptomatic COVID-19 (Infections and infestations) | NA | 1 | NA | 0 | NA
Bronchitis (Infections and infestations) | NA | 2 | NA | 1 | NA
COVID-19 (Infections and infestations) | NA | 48 | NA | 48 | NA
COVID-19 pneumonia (Infections and infestations) | NA | 1 | NA | 4 | NA
Cellulitis (Infections and infestations) | NA | 1 | NA | 0 | NA
Coronavirus infection (Infections and infestations) | NA | 1 | NA | 1 | NA
Diverticulitis (Infections and infestations) | NA | 0 | NA | 1 | NA
Empyema (Infections and infestations) | NA | 1 | NA | 0 | NA
Endocarditis (Infections and infestations) | NA | 0 | NA | 1 | NA
Herpes zoster (Infections and infestations) | NA | 0 | NA | 1 | NA
Infection parasitic (Infections and infestations) | NA | 1 | NA | 0 | NA
Kidney infection (Infections and infestations) | NA | 0 | NA | 1 | NA
Localised infection (Infections and infestations) | NA | 0 | NA | 1 | NA
Lung abscess (Infections and infestations) | NA | 1 | NA | 0 | NA
Neutropenic sepsis (Infections and infestations) | NA | 0 | NA | 2 | NA
Pneumonia (Infections and infestations) | NA | 13 | NA | 9 | NA
Pneumonia pseudomonal (Infections and infestations) | NA | 1 | NA | 0 | NA
Rectal abscess (Infections and infestations) | NA | 0 | NA | 1 | NA
Respiratory tract infection (Infections and infestations) | NA | 0 | NA | 2 | NA
Sepsis (Infections and infestations) | NA | 1 | NA | 1 | NA
Septic shock (Infections and infestations) | NA | 1 | NA | 0 | NA
Tuberculosis (Infections and infestations) | NA | 1 | NA | 0 | NA
Urinary tract infection (Infections and infestations) | NA | 1 | NA | 1 | NA
Alcohol poisoning (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA
Head injury (Injury, poisoning and procedural complications) | NA | 1 | NA | 1 | NA
Hip fracture (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA
Ligament rupture (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA
Procedural pneumothorax (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA
Radius fracture (Injury, poisoning and procedural complications) | NA | 1 | NA | 0 | NA
Spinal compression fracture (Injury, poisoning and procedural complications) | NA | 0 | NA | 1 | NA
Toxicity to various agents (Injury, poisoning and procedural complications) | NA | 0 | NA | 2 | NA
Alanine aminotransferase increased (Investigations) | NA | 0 | NA | 1 | NA
Aspartate aminotransferase increased (Investigations) | NA | 0 | NA | 1 | NA
C-reactive protein increased (Investigations) | NA | 0 | NA | 3 | NA
Electrocardiogram T wave amplitude decreased (Investigations) | NA | 0 | NA | 1 | NA
Hepatic enzyme increased (Investigations) | NA | 1 | NA | 0 | NA
Influenza A virus test positive (Investigations) | NA | 1 | NA | 0 | NA
SARS-CoV-2 test positive (Investigations) | NA | 3 | NA | 2 | NA
Hypokalaemia (Metabolism and nutrition disorders) | NA | 1 | NA | 1 | NA
Hyponatraemia (Metabolism and nutrition disorders) | NA | 1 | NA | 1 | NA
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | NA | 0 | NA | 1 | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | 2 | NA | 0 | NA
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 3 | NA
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | NA | 0 | NA | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | 1 | NA
Tenosynovitis (Musculoskeletal and connective tissue disorders) | NA | 1 | NA | 0 | NA
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 3 | NA | 1 | NA
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 0 | NA
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 0 | NA
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 2 | NA
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 0 | NA
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 2 | NA | 0 | NA
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 1 | NA
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 0 | NA
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 1 | NA | 1 | NA
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | NA | 1 | NA
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 2 | NA | 0 | NA
Altered state of consciousness (Nervous system disorders) | NA | 0 | NA | 1 | NA
Aphasia (Nervous system disorders) | NA | 0 | NA | 1 | NA
Carotid artery occlusion (Nervous system disorders) | NA | 0 | NA | 1 | NA
Cerebral infarction (Nervous system disorders) | NA | 0 | NA | 1 | NA
Cerebrovascular accident (Nervous system disorders) | NA | 4 | NA | 4 | NA
Epilepsy (Nervous system disorders) | NA | 1 | NA | 0 | NA
Generalised tonic-clonic seizure (Nervous system disorders) | NA | 1 | NA | 1 | NA
Ischaemic stroke (Nervous system disorders) | NA | 0 | NA | 1 | NA
Partial seizures (Nervous system disorders) | NA | 0 | NA | 1 | NA
Peripheral nerve palsy (Nervous system disorders) | NA | 1 | NA | 0 | NA
Syncope (Nervous system disorders) | NA | 1 | NA | 1 | NA
Thrombotic cerebral infarction (Nervous system disorders) | NA | 1 | NA | 0 | NA
Ulnar nerve palsy (Nervous system disorders) | NA | 1 | NA | 0 | NA
Schizophrenia (Psychiatric disorders) | NA | 1 | NA | 0 | NA
Calculus urinary (Renal and urinary disorders) | NA | 1 | NA | 0 | NA
Haematuria (Renal and urinary disorders) | NA | 1 | NA | 0 | NA
Hydronephrosis (Renal and urinary disorders) | NA | 0 | NA | 1 | NA
Renal colic (Renal and urinary disorders) | NA | 0 | NA | 2 | NA
Renal haemorrhage (Renal and urinary disorders) | NA | 0 | NA | 1 | NA
Urinary retention (Renal and urinary disorders) | NA | 1 | NA | 0 | NA
Benign prostatic hyperplasia (Reproductive system and breast disorders) | NA | 1 | NA | 0 | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 3 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 7 | NA | 2 | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 1 | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | 2 | NA | 0 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | NA | 3 | NA | 2 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | NA | 3 | NA | 0 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | NA | 3 | NA | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | 2 | NA | 2 | NA
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | 2 | NA | 1 | NA
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | NA | 0 | NA | 1 | NA
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | NA | 1 | NA | 0 | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 1 | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | NA | 0 | NA | 1 | NA
Embolism (Vascular disorders) | NA | 1 | NA | 0 | NA
Hypertension (Vascular disorders) | NA | 0 | NA | 1 | NA
Peripheral ischaemia (Vascular disorders) | NA | 0 | NA | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants - Pre-treatment (N=0) | Canakinumab - On-treatment (N=692) | Canakinumab - Post-treatment Follow-up (N=0) | Placebo - On-treatment (N=689) | Placebo - Post-treatment Follow-up (N=0)
Anaemia (Blood and lymphatic system disorders) | NA | 46 | NA | 50 | NA
Constipation (Gastrointestinal disorders) | NA | 34 | NA | 42 | NA
Diarrhoea (Gastrointestinal disorders) | NA | 57 | NA | 48 | NA
Nausea (Gastrointestinal disorders) | NA | 46 | NA | 51 | NA
Asthenia (General disorders) | NA | 47 | NA | 33 | NA
Fatigue (General disorders) | NA | 70 | NA | 60 | NA
Pyrexia (General disorders) | NA | 28 | NA | 43 | NA
Nasopharyngitis (Infections and infestations) | NA | 44 | NA | 33 | NA
Upper respiratory tract infection (Infections and infestations) | NA | 37 | NA | 31 | NA
Alanine aminotransferase increased (Investigations) | NA | 65 | NA | 49 | NA
Amylase increased (Investigations) | NA | 52 | NA | 51 | NA
Aspartate aminotransferase increased (Investigations) | NA | 53 | NA | 37 | NA
Lipase increased (Investigations) | NA | 47 | NA | 47 | NA
Neutrophil count decreased (Investigations) | NA | 45 | NA | 13 | NA
Weight increased (Investigations) | NA | 63 | NA | 48 | NA
White blood cell count decreased (Investigations) | NA | 35 | NA | 18 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | 74 | NA | 88 | NA
Back pain (Musculoskeletal and connective tissue disorders) | NA | 61 | NA | 56 | NA
Headache (Nervous system disorders) | NA | 31 | NA | 60 | NA
Paraesthesia (Nervous system disorders) | NA | 29 | NA | 44 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | NA | 89 | NA | 108 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 67 | NA | 50 | NA
Pruritus (Skin and subcutaneous tissue disorders) | NA | 35 | NA | 34 | NA
Hypertension (Vascular disorders) | NA | 35 | NA | 24 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03447769/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT03447769/SAP_001.pdf